CLINICAL TRIAL: NCT06588179
Title: Phase Ib/II Clinical Study of SHR-1501 Combined With SHR-2005 in the Treatment of Patients With High-Risk Non-Muscle Invasive Bladder Cancer Which is Not Completely Resectable by TURBt
Brief Title: SHR-1501 Combined With SHR-2005 for High-Risk Non-Muscle Invasive Bladder Cancer Which is Not Completely Resectable by TURBt
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, Chief Physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMIBC-NCR01
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: NMIBC
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm：SHR-1501+SHR-2005 (Experimental)
  Interventions: Drug: SHR-1501+SHR-2005

INTERVENTIONS:
Drug: SHR-1501+SHR-2005 — SHR-1501, instillation；SHR-2005, instillation

SUMMARY:
This is a single-center, single-arm, phase Ib/II study, aimed at assessing the safety and efficacy of SHR-1501 in combination with SHR-2005 as treatment for patients with high-risk non-muscle invasive bladder cancer (HR NMIBC) which is not completely resectable by transurethral resection of bladder tumor (TURBt).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, both genders
2. Previous pathological biopsy was diagnosed as high-risk NMIBC
3. Tumors cannot be completely resected by TURBT（at least 2 senior urologists assessed that the lesion area is too extensive to be completely resected）
4. Ineligible or unwilling to undergo radical cystectomy
5. TURBT was performed within 6 weeks
6. Agreed to provide cystoscopic biopsy specimens for review
7. ECOG performance status of 0-2
8. Life expectancy ≥ 2 years
9. Adequate organ function：

   1. Hematological indexes: ANC ≥1.5x10^9/L, PLT ≥100x10^9/L, Hb ≥ 90 g/L;
   2. Liver function: TBIL ≤1.5 ULN; ALT and AST≤2.5 ULN; Albumin > 3g/dL
   3. Renal function: Cr≤1.5 ULN or creatinine clearance ≥ 60 ml/min (Cockcroft-Gault formula); if proteinuria ≥++, requiring 24-hour urine protein level ≤1.0g;
   4. ECG: females QTcF ≤470ms and males ≤450ms
   5. Cardiac ultrasound: LVEF≥50%
   6. Coagulation: INR or PT ≤1.5 ULN，APTT≤1.5 ULN
10. Female or male subjects of childbearing age who have not undergo surgical sterilization shall agree to use contraceptive measures (such as intrauterine device and contraceptive pill) during the study treatment period and within 3 months after the end of the study treatment period, and both female subjects and female partners of male subjects should use highly effective contraceptive methods; the Female subjects of childbearing age who have not undergone surgical sterilization must have a negative serum HCG test result within 7 days prior to the first administration and must be non-lactating.
11. Volunteered to join the study, signed the informed consent, and had good compliance with follow-up

Exclusion Criteria:

1. Previous pathological biopsy was diagnosed with muscle-invasive bladder cancer at T2 or higher stages
2. Received any other intravesical chemotherapy treatment within 2 weeks or received any other clinical drugs within 4 weeks
3. History of allergy to any of the study drugs or study drug components
4. Upper urinary tract tumor detected by CTU or MRU during screening period or other concomitant malignant tumors within 5 years before the first administration
5. Previously received any TNFR agonist antibody therapy(such as OX40, CD27, CD357 antibodies), IL-15 agonist antibody therapy, or IL-2 agonist antibody therapy
6. Oversize surgery or severe trauma within 4 weeks before the first use of research drugs
7. Previously discontinued bladder instillation therapy due to adverse reactions such as sepsis, systemic infection, or urinary incontinence
8. Active/uncontrolled impairment of the urogenital system, kidneys, liver, gallbladder, cardiovascular system, gastrointestinal tract, nervous system, or hematopoietic system, which may lead to complications for the subject when receiving intravesical therapy and/or general anesthesia
9. A history of interstitial lung disease or non-infectious pneumonitis requiring treatment with glucocorticoids, or current presence of interstitial pneumonitis or non-infectious pneumonitis, or a history of other severe pulmonary diseases
10. A history of immunodeficiency, including HIV seropositivity, other acquired or congenital immunodeficiency diseases, a history of organ transplantation, or current use of immunosuppressants
11. History of clinically significant cardiovascular disease within 6 months before the first administration
12. Investigator-assessed concern for medication safety; severe infections requiring antibiotic, antiviral or antifungal drug control; and unexplained fever > 38.5°C within 2 weeks
13. Patient with active hepatitis B (HBeAg positive and HBV DNA≥500 IU/mL), hepatitis C (HCV antibody positive and HCV RNA higher than the detection limit of the analytical method)
14. Adverse reactions of previous anti-tumor treatment have not recovered to Grade≤1 per NCI-CTCAE v5.0
15. The presence of any other conditions that the investigator deems inappropriate to participate in this study, including serious physical or mental illness, abnormal laboratory tests, and other factors that may increase the risk of participating in the study, or interfere with the results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Phase I : Incidence of dose limiting toxicities (DLTs) | From Day 1 to Day 21
Phase I : RP2D（Recommended Phase 2 dose） | From Day 1 to 90 days after last dose
Phase I : Incidence and severity of adverse events (AEs) | From Day 1 to 90 days after last dose
Phase II : CR rate at 3 months | Approximately 2 years

SECONDARY OUTCOMES:
Phase I : CR rate at 3 months | From Day 1 to 90 days after last dose
Phase II : Incidence and severity of adverse events (AEs) | Approximately 2 years
Phase Ib/II: PR rate at 3 months | Approximately 2 years
Phase Ib/II: CR rate at 6 months and 12months | Approximately 2 years
Phase Ib/II: Duration of CR (DoR) | Approximately 2 years
Phase Ib/II: Cystectomy-Free Survival (CFS) | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided